CLINICAL TRIAL: NCT00973193
Title: Phase II Study of Preoperative Panitumumab and External Beam Radiotherapy in Patients With Locally Advanced Rectal Cancer
Brief Title: Preoperative Panitumumab and Radiotherapy in Rectal Cancer
Acronym: PrePaRad
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The intermediate analyses did not allowed to continue the clinical study.
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL-ONCO 09-001; Academic study
Record Dates: First submitted 2009-09-07; First posted 2009-09-09 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Rectal Cancer
Keywords: rectum; colorectal; cancer; adenocarcinoma; anti-EGFR; monoclonal antibodies; neoadjuvant therapy; preoperative radiotherapy
MeSH Terms: conditions — Rectal Neoplasms; Neoplasms; Adenocarcinoma | interventions — Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- panitumumab (Experimental)
  Interventions: Drug: panitumumab

INTERVENTIONS:
Drug: panitumumab — intravenous infusion of panitumumab, 6 mg per kg body weight, once every 14 days for a total of 42 days
  Other Names: Vectibix

SUMMARY:
The purpose of this study is to investigate the activity of panitumumab in combination with standard preoperative radiotherapy in locally advanced rectal cancer, followed by complete surgery and adjuvant chemotherapy.

The main hypothesis of the study is that the association of EGFR-targeting agent and radiation therapy could be as effective or even improve the rate of pathological complete tumoral response with fewer toxicities in comparison to the standard of care using chemoradiation therapy.

DETAILED DESCRIPTION:
Anti-EGFR monoclonal antibodies have radiosensitizing properties. In particular, cetuximab in combination with curative-intent radiotherapy has been reported to increase median overall survival over radiation therapy alone in locally advanced head and neck carcinoma.

Similar benefit in rectal cancer is expected. However, preliminary studies revealed that the combination of chemoradiation and cetuximab did not seem to improve the pathological tumor response. However, in the past studies, the selection of patients' population was not optimal since KRAS mutational status was not considered during recruitments.

Therefore, new trials to investigate EGFR-targeting therapies in combination with radiotherapy in wild-type KRAS patients are required.

Adjuvant chemotherapy has also shown to decrease the risk of local relapse in patients who did not receive chemotherapy during radiotherapy. In our study, since there will be no chemotherapy given during the preoperative setting, the administration of adjuvant chemotherapy postoperatively is highly recommended.

ELIGIBILITY:
Inclusion Criteria:

* ECOG Performance Status 0-1
* Histologically proven adenocarcinoma of the rectum, T3-T4 and/or N+ M0
* Wild-type KRAS
* No prior pelvic irradiation
* Normal bone marrow, hepatic, renal, cardiac functions
* No secondary malignancy
* No other active, uncontrolled disease
* Signed informed consent

Exclusion Criteria:

* KRAS mutation
* Established or suspected metastasis
* Prior pelvic irradiation
* Previous exposure to EGFR-targeting therapies
* Patients under any other investigational agent(s)
* Concurrent systemic immune therapy, chemotherapy, hormone therapy
* Drug and/or alcohol abuse
* Grade 3 to 4 allergic reaction to any of the components of the treatment
* History or presence of interstitial lung disease
* Active, uncontrolled cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | 11 weeks

SECONDARY OUTCOMES:
Safety, pathologic R0 resection, negative Circumferential Resection Margin, pathologic downstaging, tumor regression grade, quality of mesorectal excision, rate of sphincter-preservation, Disease-Free Survival, local control rate, translational research | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pascal H Machiels, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (8):
- Belgium (8):
  - Institute Jules Bordet, Brussels
  - Cliniques Universitaires Saint Luc - Université Catholique de Louvain, Brussels
  - Centre Hospitalier Notre Dame et Reine Fabiola, Charleroi
  - Centre Hospitalier de Jolimont-Lobbes, La Louvière
  - UZ Gasthuisberg, Leuven
  - Clinique et Maternité Saint Elizabeth, Namur
  - Clinique Saint Pierre, Ottignies
  - Clinique Universitaire de Mont Godinne, Yvoir